CLINICAL TRIAL: NCT06977802
Title: Design and Implementation of a Mobile App for Promoting Healthy and Sustainable Eating Among Students at the University of Parma (MAPHealthS)
Acronym: MAPHealthS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: University of Milano Bicocca (Other)
Responsible Party: Principal Investigator, Francesca Scazzina Ph.D., Associate Professor, University of Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UNIPLATE
Record Dates: First submitted 2025-03-24; First posted 2025-05-18 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Dietary Fibers; Environmental Impact; Eating Habits
Keywords: dietary fiber; mobile health; sustainable eating; RCT; university students
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group controlled trial with a 12-week duration (6-week active intervention + 6-week follow-up). Participants (n=60) are university students with low baseline fiber intake, randomly assigned to:
  Intervention group (n=30): Uses a tailored mobile app (MAPHealthS) with nutrition education, meal planning, and sustainability tips.
  Control group (n=30): No intervention.
  Key features:
  Blinding: Single-blind (outcome assessors may be blinded; participants are aware of group allocation).
  Data collection: Dietary intake (24h recalls, FFQs), biomarkers (urine/fecal), anthropometrics, and actigraphy (subgroup).
  Primary outcome: Change in daily fiber intake (g/day).
  Secondary outcomes: Diet sustainability scores, physical activity, body composition, and environmental impact.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention: Participants use the UNIPLATE mobile app, a tailored educational tool designed to promote healthy and sustainable eating.
  Features: Daily nutrition/sustainability tips, meal planning, recipe suggestions (prioritizing plant-based foods), gamified challenges, and progress tracking.
  Delivery: 6-week active phase with daily app notifications, followed by 6-week follow-up (no notifications).
  Tailoring: Content adapts to baseline food-related psychobehavioral profiles (assessed via questionnaire).
  Support: Developed with input from nutritionists, psychologists, and computer scientists (University of Parma).
  Interventions: Behavioral: Digital Nutrition Education Mobile App for Healthy and Sustainable Eating
- Control (No Intervention): Intervention: No app or active intervention; participants maintain habitual dietary behaviors.
  Monitoring: Completes identical assessments (dietary recalls, biomarkers, anthropometrics) as the intervention group.

INTERVENTIONS:
Behavioral: Digital Nutrition Education Mobile App for Healthy and Sustainable Eating — This intervention is uniquely characterized by:
  Dual Health-Sustainability Focus - Unlike most nutrition apps targeting weight loss, this integrates planetary health metrics (e.g., carbon/water footprints) alongside dietary guidance.
  Psychobehavioral Personalization - Content is tailored to four predefined user profiles (e.g., "Convenience-Seeker," "Health-Conscious") identified through baseline questionnaires, adapting messaging strategies (e.g., time-saving tips vs. environmental appeals).
  Biomarker-Validated Outcomes - Unlike apps relying solely on self-reports, efficacy is assessed via objective measures (urinary LC-MS metabolomics, fecal microbiota analysis).
  Academic Development - Designed by nutrition scientists + AI engineers (University of Parma), with recipes aligned to Mediterranean/Planetary Diet standards
  Arms: Intervention

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effectiveness of a mobile app (MAPHealthS) in promoting healthy and sustainable eating habits among university students at the University of Parma. The study aims to answer the following questions:

Does the use of the educational mobile app increase daily fiber intake among students?

Does the app improve adherence to sustainable and healthy diets (e.g., Mediterranean and Planetary diets)?

What are the effects of the app on physical activity levels, anthropometric measures, and the environmental impact of participants' diets?

Researchers will compare the intervention group (using the app) to a control group (no intervention) over a 12-week period, including a 6-week active phase and a 6-week follow-up phase.

Participants will:

Download and use the app (intervention group) or follow no intervention (control group) for 12 weeks.

Complete dietary assessments (24-hour recalls, food frequency questionnaires), provide urine and fecal samples, and undergo anthropometric measurements at multiple time points.

Wear actigraphs (a subgroup) to measure energy expenditure.

Answer questionnaires on dietary habits, physical activity, and app usability.

The study expects to see a significant increase in fiber intake (7g/day) and improved sustainability awareness among app users.

ELIGIBILITY:
Inclusion Criteria:

University students (undergraduate/graduate) at the University of Parma Age 18-29 years Italian nationality and residence in Italy Baseline fiber intake <17.7g/day (below Italian average) Ownership of an iOS/Android smartphone with internet access No current use of nutrition/health tracking apps

No self-reported:

* Chronic diseases (diabetes, metabolic disorders)
* Eating disorders
* Use of medications for hypertension/dyslipidemia
* No antibiotic/probiotic use in past 4 weeks
* Not following prescribed diets or meal plans
* Not pregnant/lactating Signed informed consent

Exclusion Criteria:

Not University students (undergraduate/graduate) at the University of Parma Not Aged 18-29 years Not Italian nationality and residence in Italy Baseline fiber intake >17.7g/day (over Italian average) Not ownership of an iOS/Android smartphone with internet access Current use of nutrition/health tracking apps

Self-reported:

* Chronic diseases (diabetes, metabolic disorders)
* Eating disorders
* Use of medications for hypertension/dyslipidemia
* Antibiotic/probiotic use in past 4 weeks
* Following prescribed diets or meal plans
* Pregnant/lactating

Not signed informed consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-04 (Actual); Primary Completion 2025-04-29 (Actual); Study Completion 2025-04-29 (Actual)

PRIMARY OUTCOMES:
Dietary Fiber Intake | Baseline (T0), after three-weeks (T1), after six-weeks (T2), after twelve-weeks (T3)
  The primary outcome measures the change in participants' daily dietary fiber intake (grams/day) after using the nutrition education mobile app for 6 weeks, compared to baseline and control group levels, using 24-hour dietary recalls and food frequency questionnaires.

SECONDARY OUTCOMES:
Planetary Diet Adherence | Baseline (T0), after twelve-weeks (T3)
  Measures improvement in adherence to a sustainable diet using the Planetary Health Diet Index (PHDI) score, calculated from the food frequency questionnaire.
  The PHDI score ranges from 0 to 150, with higher scores indicating better adherence to planetary health diet, defined by the EAT-Lancet Commission.
Mediterranean Diet Adherence | Baseline (T0), after twelve-weeks (T3)
  Assesses increased adherence to Mediterranean diet principles using the validated MedScore index. The MedScore ranges from 0 to 25, with higher scores indicating better adherence to the Mediterranean diet.
Physical Activity Levels | Baseline (T0), after three-weeks (T1), after six-weeks (T2), after twelve-weeks (T3)
  Tracks changes in weekly physical activity using the International Physical Activity Questionnaire (IPAQ). Scores are expressed in MET-minutes/week (1 MET = energy expended at rest), ranging from 0 to 10,000+, with higher scores indicating more activity. Participants are also classified into low (<600 MET-min/week), moderate (600-2999), or high (≥3000) activity levels.
Diet-Related Environmental Footprint | Baseline (T0), after three-weeks (T1), after six-weeks (T2), after twelve-weeks (T3)
  Diet-related Carbon Footprint: Measured in kg CO₂eq/day, this indicates the total greenhouse gas (GHG) emissions associated with the diet. It is assessed based on 24-hour recalls and the SU-EATABLE LIFE database, a comprehensive resource for the carbon and water footprints of food products. Lower values reflect a reduction in carbon emissions.
Diet-Related Water Footprint | Baseline (T0), after three-weeks (T1), after six-weeks (T2), after twelve-weeks (T3)
  Diet-related Water Footprint: Measured in liters/day, this indicates the total water consumption associated with the diet. It is assessed based on 24-hour recalls and the SU-EATABLE LIFE database, which provides comprehensive data on the water footprints of food products. Lower values reflect a reduction in water usage.
App Usability/Satisfaction | Twelve-weeks after enrollment (T3)
  The usability and satisfaction of the app will be assessed using the validated mHealth Satisfaction Questionnaire (a questionnaire for assessing user satisfaction with mobile health apps, developed by Melin et al., 2020, using rasch measurement theory. In addition to the these questions, several case-specific questions were added to tailor the assessment to the app's unique features. Participants will also be asked open-ended questions to gather qualitative feedback on their experience. The scale uses Likert-type responses (e.g., 1 = Strongly Disagree to 5 = Strongly Agree), and the responses will be analyzed to identify patterns in user satisfaction and usability. Higher scores reflect greater satisfaction and perceived usability.
Biomarker Validation | Baseline (T0), after three-weeks (T1), after six-weeks (T2)
  Validates dietary changes through:
  Urinary liquid chromatography-mass spectrometry (LC-MS) metabolomics (polyphenol metabolites)
  Fecal microbiota analysis (16S rRNA sequencing)

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Scazzina, Principal Investigator — Università di Parma
Locations (1):
- Plesso Biotecnologico Integrato, Parma, PR, Italy

IPD SHARING:
Plan to Share IPD: Undecided